CLINICAL TRIAL: NCT04458714
Title: Carbon Dioxide Versus Iodine Contrast Medium for Endovascular Revascularization of Aortoiliac Occlusive Disease: A Two Center Randomized Controlled Trial
Brief Title: Carbon Dioxide Versus Iodine Contrast for Endovascular Revascularization of Aortoiliac Occlusive Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Amro Elboushi, associate professorof vascular surgery, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: zu-irb#6036/16-3-2015
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Aortoiliac Occlusive Disease
Keywords: CO2 angiography; angioplasty; aortoiliac occlusive disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients who agreed were asked to sign an informed consent. After patient data input was done, randomization was computer generated in the vascular surgery department in Zagazig university hospitals. Computer generated random numbers were created with the use of randomly permuted blocks with two block sizes; after which they were secured in consecutive numbered envelopes and group allocation was independent of time and person delivering the treatment. Single blinding was used to recruit the patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CO2 group (treatment arm) (Active Comparator): This arm included 32 patients who were randomized for using CO2 as the contrast medium for aortoiliac angiolplasty.
  Interventions: Procedure: Aortoiliac angioplasty
- ICM group (control arm) (Active Comparator): This arm involved 32 patients who were randomized for using iodine contrast medium (ICM) for aortoiliac angiolplasty.
  Interventions: Procedure: Aortoiliac angioplasty

INTERVENTIONS:
Procedure: Aortoiliac angioplasty — In the CO2 arm we used manual injection of CO2 from a medicinal CO2 cylinder connected to a particle filter. Under water aspiration was used to prevent air contamination. Using a twenty mls syringe the required amount of CO2was aspirated using a three way tap and was followed my aspirating 3mls of saline to provide a fluid barrier. In the ICM arm the injection of contrast was done using 10-ml syringes with 5 mls of iodinated contrast media and 5 mls of saline solution per injection. The ICM used in all cases was Omnipaque 300 (Iohexol), a nonionic low osmolar contrast commonly in use in both hospitals.

SUMMARY:
From July 2015 to July 2018, 64 patients with aortoiliac occlusive disease who were eligible for endovascular treatment and lacked contraindications to either iodine contrast or carbon dioxide (CO2) were randomized into the carbon dioxide CO2 group(32) or iodine contrast medium(ICM) group(32) were subjected to aortoiliac angioplasty. The primary outcome was the quality of image as the sole contrast agent used in interventions. The secondary outcomes were technical success rate and the safety of procedure.

DETAILED DESCRIPTION:
Sampling The sample size was calculated by the intuitional review board statistician using open epi based on the RCT done by Mendes et al. Power of study as set at 80% and confidence interval set at 95%. The sample size was calculated to be 64 cases, 32 in each group.

Randomization All patients who qualified for the inclusion and exclusion criteria were offered to participate in the trial after explaining all the details involved with the potential benefits and risks of both contrast mediums. Patients who agreed were asked to sign an informed consent. After patient data input was done, randomization was computer generated in the vascular surgery department in Zagazig university hospitals. Computer generated random numbers were created with the use of randomly permuted blocks with two block sizes; after which they were secured in consecutive numbered envelopes and group allocation was independent of time and person delivering the treatment. Single blinding was used to recruit the patients. The patients were randomized into the following two arms: a CO2 group (treatment arm) and an ICM group (control arm) according to the contrast medium selected for the intervention. Group I included 32 patients who were randomized for using CO2 as the contrast medium. Group II: involved 32 patients who were randomized for using iodine contrast medium (ICM).

Postoperative assessment and follow-up The endovascular equipment used in each intervention and the volumes of contrast used were accurately documented for analysis. Immediately after the operation all patients in both arms received intravenous fluids pre and post intervention following a local guideline for renal protection.¬ Patients were discharged the next day and outpatient renal functions were repeated 3 days post procedure, 1 week and 1 month. We analyzed creatinine levels between the two groups during the pre- and post-operative periods. Any elevation of serum creatinine (Scr) of more than 25% or ≥0.5 mg/dl is defined as contrast induced nephropathy (CIN). Patients were followed up for 1 year. One patient from the CO2 group decided to withdraw from the trial during the follow up period and was excluded from the follow up analysis.

Imaging from all cases were analyzed on conclusion of the study. The images were reviewed by two independent observers (radiologists with > 5 years of experience in performing endovascular procedures) blinded to treatment arm. Image quality was assessed using Likert rating scale ranging from 1 (very poor) to 5 (very good) for each image.18 A score of 1 was defined as poor quality with loss of delineation of the vessel. A score of 2 was considered below average with poor delineation of the vessel, a score of 3 is for average quality image and medium delineation of the vessel, a score of 4 was considered good quality with clear delineation of the vessel and a score of 5 was considered very good quality with very clear delineation of the vessel.

ELIGIBILITY:
Inclusion Criteria:

* Patients with aortoiliac arteries atherosclerotic disease (with arterial atherosclerotic disease classified as Trans-Atlantic Inter-Society Consensus (TASC) A, B and C, (classified by CT angiography)
* Patients with good distal runoff
* Patients suitable for either types of contrast ICM or CO2 (No history of allergy to contrast and normal kidney functions)

Exclusion Criteria:

* Patients with TASC D aortoiliac lesions
* Patients requiring femoral endartectomy
* Patient s with significant multilevel distal disease
* Patients suffering from severe chronic obstructive lung disease, chronic kidney failure, heart failure, or pregnancy.
* Patients younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
quality of image as the sole contrast agent to perform the needed interventions: Likert rating scale | on conclusion of patient recruitment , image quality was aseessed within 12 weeks
  Imaging from all cases were analyzed on conclusion of the study. The images were reviewed by two independent observers (radiologists with > 5 years of experience in performing endovascular procedures) blinded to treatment arm. Image quality was assessed using Likert rating scale ranging from 1 (very poor) to 5 (very good) for each image.

SECONDARY OUTCOMES:
technical success rate | immediate post operative
  surgical results with completion of the intended procedure.
Incidence of Procedure-related complications . | 1year follow up
  defined as the freedom from procedural complications (Procedure-related complications were the incidence of cardiac death, myocardial infarction, stroke, major amputation, non-occlusive mesenteric ischemia, extended hospitalization (> 24 hours) as a consequence of CO2-guided treatment, hematomas, pseudo-aneurysms, perforations, contrast induced nephropathy (CIN), target lesion revascularization and postoperative death within 3 months of surgery,)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Almeida Mendes C, de Arruda Martins A, Teivelis MP, Kuzniec S, Nishinari K, Krutman M, Halpern H, Wolosker N. Carbon dioxide is a cost-effective contrast medium to guide revascularization of TASC A and TASC B femoropopliteal occlusive disease. Ann Vasc Surg. 2014 Aug;28(6):1473-8. doi: 10.1016/j.avsg.2014.03.021. Epub 2014 Apr 3. PMID 24704050
- [Background] Fujihara M, Kawasaki D, Shintani Y, Fukunaga M, Nakama T, Koshida R, Higashimori A, Yokoi Y; CO2 Angiography Registry Investigators. Endovascular therapy by CO2 angiography to prevent contrast-induced nephropathy in patients with chronic kidney disease: a prospective multicenter trial of CO2 angiography registry. Catheter Cardiovasc Interv. 2015 Apr;85(5):870-7. doi: 10.1002/ccd.25722. Epub 2014 Nov 21. PMID 25380326
- [Background] Sharafuddin MJ, Marjan AE. Current status of carbon dioxide angiography. J Vasc Surg. 2017 Aug;66(2):618-637. doi: 10.1016/j.jvs.2017.03.446. PMID 28735955